CLINICAL TRIAL: NCT03158415
Title: Parents of Young Adults With Type 1 Diabetes: An Exploratory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB201700810; 13177 (Other: University of Florida)
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Type1diabetes; Parents
Keywords: mHealth

STUDY DESIGN:
Intervention Model Description: Mixed Methods Exploratory Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parents of Young Adults with T1D (Experimental): Parents of young adults ages 18 to 25 years with type 1 diabetes who are transitioning to independence. During six weeks, participants will receive a reminder via text and/or email twice per week to invite them to view diabetes education materials on the study's mobile website, T1DToolkit.org. Topics on this website include, among others, Caregiver Burnout; Your Child is Now an Adult; Sharing Responsibility; Sources of Support; Common Fears for Parents of Young Adults; and Your Child, Your Child's Doctor, and You.
  Interventions: Behavioral: T1DToolkit.org mobile diabetes education

INTERVENTIONS:
Behavioral: T1DToolkit.org mobile diabetes education — Participants will receive a reminder via text and/or email twice per week to invite them to view diabetes education materials on the study's mobile website, T1DToolkit.org. Topics on this website include, among others, Caregiver Burnout; Your Child is Now an Adult; Sharing Responsibility; Sources of Support; Common Fears for Parents of Young Adults; and Your Child, Your Child's Doctor, and You.
  Six weeks after enrollment, participants will complete the Modified Diabetes Distress Scale: Parents of Young Adults.

SUMMARY:
The purpose of this mixed-methods study is to explore the lived experience of parents of young adults ages 18 to 25 years with type 1 diabetes who are transitioning to independence, and to test the preliminary efficacy of a mobile education program to reduce parental distress.

DETAILED DESCRIPTION:
As young adults with T1D navigate the transition process to independence, they often do so in partnership with their parents, who are tasked with providing support and guidance. At this time, however, no structured education program exists for these parents. In addition, little is known about their learning needs, levels of distress, and readiness to provide appropriate guidance for their emerging adult children. This represents a gap in the literature and an opportunity to undertake exploratory research to learn more about this population so that meaningful education and support can be provided.

Aim 1. To describe the lived experience and diabetes-specific educational needs of parents of young adults with type 1 diabetes who are transitioning to independence.

Aim 2. To measure the effect of a mobile diabetes education program on diabetes distress levels of parents of young adults ages 18 to 25 years who are transitioning to independence.

ELIGIBILITY:
Inclusion Criteria:

* (1) Ability to read and speak English
* (2) parent of a child aged ≥18 years and ≤25 years with a diagnosis with T1D
* (3) must have access to a smartphone or tablet or laptop/desktop computer with internet access.

Exclusion Criteria:

* (1) Significant medical comorbidity in the participant that could, in the opinion of the PI, affect participant's capacity to complete study follow up;
* (2) inability to read and speak English.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
Lived experience | 1 week
  The transcripts of the semi-structured interviews will be coded and analyzed using qualitative data content analysis to describe the the lived experience and diabetes-specific educational needs of parents of young adults with type 1 diabetes who are transitioning to independence.

SECONDARY OUTCOMES:
Diabetes Distress | 6 weeks
  The Modified Diabetes Distress Scale will be used pre- and post-intervention to measure the effect of a brief mobile diabetes education program on diabetes distress levels of parents of young adults ages 18 to 25 years who are transitioning to independence. Higher scores on the Distress Scale indicate higher levels of distress.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Albanese-O'Neill, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No